CLINICAL TRIAL: NCT07247656
Title: Comparison of Empagliflozin- Linagliptin With Empagliflozin- Metformin Combination Therapy in Reduction of Body Weight in Type 2 Diabetes Mellitus
Brief Title: The Efficacy and Safety of Empagliflozin - Linagliptin and Empagliflozin- Metformin Therapy in Reduction of Body Weight in Type 2 Diabetic Patients .
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bahria University (Other)
Responsible Party: Principal Investigator, Dr. Nabila Rafi, MBBS , M.PHIL PHARMACOLOGY, Bahria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ERC 105/2022
Record Dates: First submitted 2025-09-17; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Diabete Mellitus
Keywords: liver profile; BMI; Waist to Hip Ratio; Renal Function tests; HBA1C
MeSH Terms: conditions — Diabetes Mellitus | interventions — empagliflozin; Linagliptin; Metformin

STUDY DESIGN:
Intervention Model Description: The patients was be divided two groups on the basis of their treatment option; group A Empagliflozin with Linagliptin group B Empagliflozin with Metformin
  The study was be ethically approved by the Bahria University ethical review committee (BUMDC). Informed consent was taken before initiating the clinical trial in male and female diabetic patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group B received Empagliflozin with Linagliptin (Active Comparator): Empagliflozin 10 mg, along with Tab Linagliptin 5mg.
  Interventions: Drug: (Empagliflozin 10 mg+ Tab Linagliptin 5mg)
- Group A received Empagliflozin with Metformin (Active Comparator): Tab Empagliflozin 10 mg once daily, along with combination of Tab Metformin 500 mg
  Interventions: Drug: Tab Empagliflozin 10 mg + Tab Metformin 500 mg

INTERVENTIONS:
Drug: (Empagliflozin 10 mg+ Tab Linagliptin 5mg) — (Empagliflozin 10 mg+ Tab Linagliptin 5mg)was given once Orally daily
  Other Names: Diampa LT (10/5 ) MG; Xenglu- Lin (10 / 5 ) MG; Empaa L ( 10 / 5 ) MG
  Arms: Group B received Empagliflozin with Linagliptin
Drug: Tab Empagliflozin 10 mg + Tab Metformin 500 mg — Tab Empagliflozin 10 mg once daily, along with combination of Tab Metformin 500 mg
  Other Names: Xenglu - Met XR ( 10 / 500 ) MG
  Arms: Group A received Empagliflozin with Metformin

SUMMARY:
The goal of this clinical trial is - Comparison of Empagliflozin - Linagliptin with Empagliflozin - Metformin combination therapy in reduction of body weight in T2DM Patients and it included 200 diabetic subjects with total study period of 12 weeks and individual study period of 4 weeks .

DETAILED DESCRIPTION:
The goal of this clinical trial is to evaluate the safety and efficacy of both the drugs combination in evaluating weight loss and glycemic parameters .

SPSS version 25 will be used to generate the descriptive statistics. Frequency and percentage figures will be used to represent the qualitative factors.

The comparison will be done between male of group A with male of group B and female of group A with female of group B.

ELIGIBILITY:
Inclusion Criteria:

* • Diabetic men and women of age 40-70 yrs.

  * HBA1C -(6.5-9 )percent
  * All diabetic patients were BMI ≥25kg/m2
  * Patient took metformin ≥1000mg/day for ≥ 3 months with uncontrolled DM

Exclusion Criteria:

* Male and female type 1 diabetic patients with BMI <25

  * Diabetic patient taking oral medicine other than metformin for last 12 weeks
  * Subjects with creatinine >1.5mg/dl
  * Pregnant or Lactating Women
  * Co-morbidities -
  * CLD
  * Cancer patient

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Overall improvement in Fasting Blood Glucose | 12 weeks
  Fasting Blood glucose ( mg / dl ) was measured using Glucometer
Overall change in Body Mass Index ( kg/m2) | 12 weeks
  Body Mass Index ( kg/m2) was recorded using weighing balance and measuring tape .
Overall improvement in Random Blood Glucose | 12 weeks
  Random Blood Glucose was measured in mg/dl using Glucometer
Over all improvement in Glycated Hemoglobin ( HbA1c) | 12 weeks
  Blood sample was taken to assess HbA1c
Overall change in Waist to Hip Ratio | 12 weeks
  Measuring tape was used to measure
Overall change in Waist Circumference | 12 weeks
  Was measured in inches using measuring tape

SECONDARY OUTCOMES:
To observe adverse effects in treatment groups | 12 weeks
  1. To evaluate any incidence of Hypoglycemic events during study period
  2. To evaluate any incidence of Glycosuria during study period

CONTACTS AND LOCATIONS:
Overall Officials: NABILA RAFI, Principal Investigator — DOCTOR
Locations (1):
- Bahria University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD data will be shared
Supporting Information: Study Protocol
Time Frame: 1 year after article publication
Access Criteria: Access to all
URL: https://www.bahria.edu.pk/bukc